CLINICAL TRIAL: NCT03871686
Title: Improving Well-being Among Young Adult Survivors of Childhood Brain Tumor: A Randomized Controlled Trial of a Brief Internet-based Behavioral Activation Program
Brief Title: Promotion of Well-being of Young Adult Brain Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0006; A177800 (Other: UW, Madison); EDUC/REHAB PSYC&SP ED (Other: UW, Madison)
Record Dates: First submitted 2019-01-19; First posted 2019-03-12 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Brain Tumor, Pediatric
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: The experimental group will take a 4-session Internet-based behavioral activation intervention and the control group will receive no treatment and may continue services as usual as provided by the Children's Brain Tumor Foundation.
Masking Description: Investigators and participants will know which arm of the study participants are randomly assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will be asked to complete a brief online program over a 4 to 8-week period. Each week participants will be asked to complete one session of the program online. There are four sessions.
  Interventions: Behavioral: Brief Internet-based Behavioral Activation Intervention
- Control Group (No Intervention): Participants will receive no intervention from the investigators. Participants may continue services as usual as provided by Children's Brain Tumor Foundation.

INTERVENTIONS:
Behavioral: Brief Internet-based Behavioral Activation Intervention — A brief Internet-based behavioral activation intervention consisting of 4 sessions.
  Other Names: Taking Action and Making Commitment: A Well-being Prorgram
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an Internet-based, behavioral activation intervention to promote well-being in a young adult survivors of childhood brain tumor.

DETAILED DESCRIPTION:
Participants will be recruited through the Children's Brain Tumor Foundation who will share the study announcement with their young adult members and social media. Eligible participants will complete a baseline battery survey via Qualtrics. The investigators will recruit 120 participants. The survey will take approximately 30 minutes to complete. Participants will be randomly assigned to an experimental group or control group. The experimental group will take an Internet-based behavioral activation intervention. The intervention has four modules and will be administered via Qualtrics. A link to each module will be sent to the participants via e-mail. Participants will have one week to complete each module. Once a participant completes a module, the next module link will be sent after 3 days. A reminder will be sent at 7 days and 10 days until the module is complete. Each module will take approximately 30 minutes to complete. The experimental group may continue to receive services as usual from the Children's Brain Tumor Foundation. The control group will continue to receive services as usual from the Children's Brain Tumor Foundation. The control group will have an opportunity to take the intervention once data collection is complete. Both groups will be asked to complete a battery of surveys at the end of the intervention and intermittently over a 3-month period.

ELIGIBILITY:
Inclusion Criteria:

* History of childhood brain tumor
* Ages of 18 and 30 years.
* Have regular access to the Internet
* Provide an e-mail address

Exclusion Criteria:

* Those that do not meet the inclusion criteria.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline PERMA-Profiler score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  The PERMA-Profiler is a general measure of well-being (Butler & Kern, 2016). The PERMA-Profiler measures Seligman's (2011) five pillars of well-being: positive emotion, engagement, relationships, meaning, and accomplishment. The measure consists of 23 items, including three items for each domain. The health, negative emotion, loneliness, and overall happiness items act as filler questions and provide more information. Items are rated on an 11-point Likert scale ranging from 0 (never) to 10 (always), or 0 (not at all) to 10 (completely). Scores are calculated as the average of the items comprising each factor. Butler and Kern (2016) suggested that the multidimensional structure be retained, rather than condensing responses; however, a single well-being score may provide a global indication of well-being. Therefore, for the current study, total scores for each subscale will be calculated as well as the total scores. Change from baseline total score will be assessed.

SECONDARY OUTCOMES:
Change from baseline World Health Organization-Disability Assessment Schedule 2.0 score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  Measures overall health, functioning, and disability. Total scores range from 0 to 24. Scores are summed with higher scores indicating greater functional disability severity.
Change from baseline Life Satisfaction Scale (LiSat-9) score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  To measure satisfaction with life, the Life Satisfaction Questionnaire (LiSat-9; Fugl-Meyer et al., 1991) will be included. The LiSat-9 has 9 items; including one general life satisfaction item. There 8 are domain-specific items for vocational situation, financial situation, leisure, contact friends, sexual life, activities of daily living, family life, and partnership relationship. Items are rated on an Likert scale ranging from 1 (very dissatisfying) to 6 (very satisfying). Scoring consists of calculating the mean score. Higher scores indicate greater satisfaction with life.
Change in baseline Perceived Stress Scale score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  To measure perceived stress, the Perceived Stress Scale (PSS; Cohen & Williamson, 1988) will be used. The PSS is a widely used 10-item scale in which respondents rate how stressful (unpredictable, uncontrollable, and overloaded) they perceive their lives to have been within the past month. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Scoring consists of calculating the mean score. Higher scores indicate greater perceived stress.
Change in baseline Acceptance and Action Questionnaire (AAQ-II) score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  The Acceptance and Action Questionnaire (AAQ-II) (Bond et al., 2011) consists of seven items to be answered on a scale of 1 (never true) to 7 (always true). The AAQ-II measures participants' willingness to live in accordance with their values, in contact with negative private events, and acceptance of these events. A higher total score indicates a higher level of psychological flexibility, that is higher acceptance and less experiential avoidance. Total mean score will be calculated.
Change in baseline Behavioral Activation for Depression Scale (BADS-9) score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  The Behavioral Activation for Depression Scale- Short Form (BADS-9) is a 9-item scale with scores ranging from 0 to 54, with high scores representing higher activation. Total mean scores will be calculated.
Change in baseline Cognitive-Behavioral Social Self-Efficacy Scale score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  The Cognitive-Behavioral Social Self-Efficacy Scale is an 18-item measure of perceived social self-efficacy. Item scores range from 1 (not confident at all) to 5 (very confident. Total scores range from 18 to 90, with higher scores representing greater perceived social self-efficacy. Total mean scores will be calculated.
Change in baseline Vocational Outcomes Expectancy Scale score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  The Vocational Outcome Expectancy Scale (VOES) measures outcome expectancy related to employment. It is an 11-item scale with item scores ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 11 to 55, with higher scores representing a greater expectation of attaining positive employment outcomes (i.e., obtaining or retaining employment). Total mean scores will be calculated.
Change in baseline Perceived Barrier Scale score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  The Perceived Career Barriers measure was developed to identify barriers to career development and employment of young adult survivors of pediatric brain tumors (Strauser et al., 2018). The 12-item measure uses an 11-point Likert Scale (0-10) with 0 being (not a barrier) and 10 being a (major barrier). A midpoint label of (somewhat of a barrier) is utilized. Total scores range from 0 to 110, with higher scores indicating greater perceived career barriers.
Change in baseline General Self-Efficacy Scale score at 2 weeks and 3 months | At baseline; 2 weeks and 3 months after completing the intervention.
  The General Self-Efficacy Scale (GSES) is a measure of general self-efficacy. It is a 10-item measure with item scores ranging from 1 (not true at all) to 4 (exactly true). Total scores range between 10 and 40, with a higher score indicating more self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Tansey, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Children's Brain Tumor Foundation, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No